CLINICAL TRIAL: NCT05842772
Title: Feasibility Testing a shareD dEciSIon Making Intervention for People With Kidney failuRE (DESIRE), Their Relatives, and the Health Professionals in Kidney Services: a Pilot Randomized Controlled Trial Study Protocol
Brief Title: Feasibility Testing a shareD dEciSIon Making Intervention for People With Kidney failuRE, Their Relatives, and the Health Professionals in Kidney Services: a Pilot Randomized Controlled Trial Study Protocol
Acronym: DESIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PilotRCT_LEB
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-02

CONDITIONS: Kidney Failure; End of Life
Keywords: Shared decision making; Patient decision aid
MeSH Terms: conditions — Renal Insufficiency; Death

STUDY DESIGN:
Intervention Model Description: The DESIRE trial is designed as a pragmatic, pilot, randomized, controlled, non-blinded multicenter superiority trial with two parallel groups will test the acceptability and feasibility of the intervention on patients, relatives, and health professionals.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independant research assistant will type the answers into Excel. The study principal investigator will conduct the data analyses and will be blinded to the identity of the participants only knowing them by their unique number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The DESIRE intervention which includes training of health professionals, a conversation with patients and their relatives, and a patient decision aid.
  Interventions: Other: Shared decision making intervention for patients with kidney failure when planning end-of-life care
- Control group (Active Comparator): Usual care
  Interventions: Other: Shared decision making intervention for patients with kidney failure when planning end-of-life care

INTERVENTIONS:
Other: Shared decision making intervention for patients with kidney failure when planning end-of-life care — Testing a shared decision making intervention and a patient decision aid for patients with kidney failure, their relatives, and the health professionals.

SUMMARY:
The aim of this research is to test the acceptability and feasibility of a shared decision making intervention and a patient decision aid to support patients with kidney failure, relatives, and health professionals in planning and deciding about end-of-life care together.

DETAILED DESCRIPTION:
The objectives of this study is to pilot test an intervention aiming to accomplish shared decision making when deciding about end-of-life care preferences in people with kidney failure. The intervention consists of shared decision making consultations for adults with kidney failure their relatives and contact health professionals regarding end-of-life care planning supported by a patient decision aid. We will evaluate how adults, relatives and, health professionals implements the intervention and if the intervention is acceptable to the different stakeholders. The research question will investigate if the adults, relatives, and health professionals are experiencing the intervention as shared decision making and if they feel involved in the decision making process.

The DESIRE trial is designed as a pragmatic, pilot, randomized, controlled, non-blinded multicenter superiority trial with two parallel groups will test the acceptability and feasibility of the intervention on patients, relatives, and health professionals. Randomization will be performed as block randomization with a 1:1 allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adults with kidney failure on haemodialysis, peritoneal dialysis, or on conservative kidney management and their relatives will be considered for participation. Inclusion criteria will be adults ≥75 years of age, with an estimated glomerular filtration rate <15, and not suited for a kidney transplant.

Exclusion Criteria:

* Adults who are cognitively unable to participate will be excluded from the research.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
change in the patient's palliative care needs | Through study completion, an average of 6 months
  The primary outcome will be the change in the adults' palliative needs, as measured using the Integrated Palliative Outcome Score (IPOS)-Renal patient version questionnaire

SECONDARY OUTCOMES:
Participants and relatives' experiences of shared decision making and health professionals' conduction of shared decision making are secondary outcomes. | Through study completion, an average of 6 months
  Participants and relatives' experiences of shared decision making, as measured using the Patient Experience of Shared Decision Making (SHARED) tool and healthprofessionals' conduction of shared decision making, as measured using the Decision Support Analysis Tool (DSAT-10) are secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Engelbrecht Buur, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buur LE, Bekker HL, Sondergaard H, Kannegaard M, Madsen JK, Khatir DS, Finderup J. Feasibility and acceptability of the ShareD dEciSIon making for patients with kidney failuRE to improve end-of-life care intervention: A pilot multicentre randomised controlled trial. Int J Nurs Stud Adv. 2024 Aug 5;7:100231. doi: 10.1016/j.ijnsa.2024.100231. eCollection 2024 Dec. PMID 39221228